CLINICAL TRIAL: NCT01785823
Title: The Efficacy of the Time-scheduled Decremental Continuous Infusion of Fentanyl for Postoperative Patient-controlled Analgesia After Total Intravenous Anesthesia
Brief Title: Fentanyl Background Infusion for Acute Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-DEV-DE1-11-288
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Analgesia Disorder
Keywords: analgesia; fentanyl; total intravenous anesthesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FX2-2-2 (Experimental): Their background infusions of fentanyl diluent (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at the fixed-rate of 2 ml/hr until the postoperative 24 hr
  Interventions: Other: D6-4-2; Other: D8-4-2
- D6-4-2 (Active Comparator): Their background infusions of fentanyl diluent (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at the decremental rates of 6.0 ml/hr (D6-4-2) during 1 hr, 4.0 ml/hr during 1~3 hr and 2.0 ml/hr during 3~24 hr,
  Interventions: Other: FX2-2-2; Other: D8-4-2
- D8-4-2 (Active Comparator): Their background infusions of fentanyl diluent (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at at the decremental rates of 8.0 ml/hr (D8-4-2) during 1 hr, 4.0 ml/hr during 1~3 hr and 2.0 ml/hr during 3~24 hr,
  Interventions: Other: FX2-2-2; Other: D6-4-2

INTERVENTIONS:
Other: FX2-2-2 — Their background infusions of fentanyl diluent (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at the fixed-rate of 2 ml/hr until the postoperative 24 hr (FX2-2-2), or at the decremental rates of 6.0 ml/hr (D6-4-2) and 8.0 ml/hr (D8-4-2) during 1 hr, 4.0 ml/hr during 1~3 hr and 2.0 ml/hr during 3~24 hr, postoperatively. The visual analogue scores (VAS), the incidence of inadequate analgesia, the frequency of intervention of PCA, and side effects were evaluated.
  Other Names: decremental PCA
  Arms: D6-4-2; D8-4-2
Other: D6-4-2 — Their background infusions of fentanyl diluent (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at the fixed-rate of 2 ml/hr until the postoperative 24 hr (FX2-2-2), or at the decremental rates of 6.0 ml/hr (D6-4-2) and 8.0 ml/hr (D8-4-2) during 1 hr, 4.0 ml/hr during 1~3 hr and 2.0 ml/hr during 3~24 hr, postoperatively. The visual analogue scores (VAS), the incidence of inadequate analgesia, the frequency of intervention of PCA, and side effects were evaluated.
  Other Names: decremantl PCA 6-4-2
  Arms: D8-4-2; FX2-2-2
Other: D8-4-2 — Their background infusions of fentanyl diluent (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at the fixed-rate of 2 ml/hr until the postoperative 24 hr (FX2-2-2), or at the decremental rates of 6.0 ml/hr (D6-4-2) and 8.0 ml/hr (D8-4-2) during 1 hr, 4.0 ml/hr during 1~3 hr and 2.0 ml/hr during 3~24 hr, postoperatively. The visual analogue scores (VAS), the incidence of inadequate analgesia, the frequency of intervention of PCA, and side effects were evaluated.
  Other Names: decremental PCA 8-4-2
  Arms: D6-4-2; FX2-2-2

SUMMARY:
We investigated the efficacy and the safety of the pharmacokinetic model-based patient-controlled analgesia (PCA) regimens of fentanyl for postoperative analgesia after total intravenous anesthesia (TIVA).

DETAILED DESCRIPTION:
Infusions of fentanyl (2 ml/hr of diluent was equivalent with 0.5 μg/kg/hr of fentanyl) were maintained at the fixed-rate of 2 ml/hr until the postoperative 24 hr, or at the decremental rates of 6.0 ml/hr or 8.0 ml/hr during 1 hr, 4.0 ml/hr during 1~3 hr and 2.0 ml/hr during 3~24 hr, postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients who had undergone patient-controlled analgesia (PCA) after hysterectomy

Exclusion Criteria:

* neurologic disorders
* psychiatric disorders
* renal or hepatic disorders

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
visual analogue scores (VAS) | until post-operative 24 hrs
  The assessments of analgesia and patient condition were performed at the time points of immediate post-operative periods (1, 15, 30, 45, and 60 min) and post-operative 2, 3, 4, 6, 12 and 24 hr.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, M.D, Principal Investigator — Ajou University
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeongki-do, South Korea